CLINICAL TRIAL: NCT02095977
Title: Insulation Failure in St. Jude Riata Leads: Screening and Predicting Impending Lead Failure
Brief Title: Insulation Failure in St. Jude Riata Leads
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hartford Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: ZWEI003872
Record Dates: First submitted 2014-01-28; First posted 2014-03-26 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Implanted With Any Currently (and Any Future) FDA-approved Medtronic ICD or CRT Device; to Which is Attached a St. Jude Riata Lead
Keywords: St. Jude Riata lead failure; implantable cardioverter-defibrillator (ICD); externalized conductors; ventricular tachyarrythmia; electrophysiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- participants (Other): all subjects meeting inclusion and none of exclusion criteria
  Interventions: Procedure: fluoroscopy; Procedure: synchronized high-voltage shock; Procedure: Holter monitor

INTERVENTIONS:
Procedure: fluoroscopy — Fluoroscopic evaluation of three different views (left anterior oblique, right anterior oblique and anterior/posterior) and magnification will be performed to check for externalized cables at 15 frames per second using the best visualized angle per screening electrophysiologist.
Procedure: synchronized high-voltage shock — If fluoroscopic evaluation shows externalized conductors or if patient is deemed high-risk, the patient will be consented for synchronized high voltage shock through his/her device. This will be done in the non-invasive electrophysiology lab with conscious sedation as is done during defibrillation threshold testing.
  For patients undergoing a generator (ICD) change as part of standard of care, performance of synchronized, high-voltage shock will be performed at the discretion of the electrophysiologist.
Procedure: Holter monitor — Participants will be given a 24-hour Holter monitor at baseline and once annually, and will be followed at least every three months throughout the study. Participants who are found to have an electrical abnormality at any point during the study may be given a 24-hour Holter monitor if it is believed that this procedure will provide clinically useful information regarding the integrity of the lead.

SUMMARY:
A recent study evaluated the Manufacturer and User Facility Device Experience (MAUDE) database, which contains reports of adverse events involving medical devices6,9. The FDA updates the database every two months. A total of 107 Riata leads with reported inside-out insulation breaks were found, of which 105 were available for analysis. The average age of the leads was 62.1+/-18.6 months. A total of 226 insulation defects were found with 143 inside-out insulation abrasions. Twenty-eight of the 105 leads (26.7%) had inside-out insulation defects underneath one or more of the high voltage-shocking coil. Of these, 23 were 8F and five were 7F Riata ST leads. Exposed cables or conductors were present in 32 leads and six leads had melted cables, presumably due to one or more high voltage shocks. 22 of the 43 leads assessed (51.2%) also had abraded ETFE cable coating exposing the conductor. Noise and other sensing issues were the most common signs of failure. Seven leads were found to have externalized cables and five exhibited electrical abnormalities. 31 patients (29.5%) experienced inappropriate shocks of which 41% had abraded cables.

A critical decision facing physicians is how to screen and manage patients who are found to have externalized cables. Externalized cables on fluoroscopy may precede any electrical abnormalities. Also noise may not be detected on all ICD models. A recent case report suggested that changes in lead parameters might be transient and may be missed. The lead may function normally as the high-voltage and pace-sense cables are covered with ETFE, which serves as the second insulating barrier. As this is a very thin layer (0.0015 inches) the reliability of this to withstand a high-energy shock is unknown. This may lead to failure of appropriate therapy for life threatening arrhythmias.

The aim of this study is to screen patients with ICD leads that potentially could have multiple different failure mechanisms, including inside-out insulation breaks, to develop a novel new algorithm and methods to detect these defects, thereby enabling physicians to prevent complications from failure of these leads.

It is hypothesized that current monitoring tools are insufficient for detecting the sometimes transient electrical failures of the Riata family of leads, and that additional device diagnostic information in combination with fluoroscopy may improve detection of electrical failures.

DETAILED DESCRIPTION:
A recent study evaluated the Manufacturer and User Facility Device Experience (MAUDE) database, which contains reports of adverse events involving medical devices6,9. The FDA updates the database every two months. A total of 107 Riata leads with reported inside-out insulation breaks were found, of which 105 were available for analysis. The average age of the leads was 62.1+/-18.6 months. A total of 226 insulation defects were found with 143 inside-out insulation abrasions. Twenty-eight of the 105 leads (26.7%) had inside-out insulation defects underneath one or more of the high voltage-shocking coil. Of these, 23 were 8F and five were 7F Riata ST leads. Exposed cables or conductors were present in 32 leads and six leads had melted cables, presumably due to one or more high voltage shocks. 22 of the 43 leads assessed (51.2%) also had abraded ETFE cable coating exposing the conductor. Noise and other sensing issues were the most common signs of failure. Seven leads were found to have externalized cables and five exhibited electrical abnormalities. 31 patients (29.5%) experienced inappropriate shocks of which 41% had abraded cables.

A critical decision facing physicians is how to screen and manage patients who are found to have externalized cables. Externalized cables on fluoroscopy may precede any electrical abnormalities. Also noise may not be detected on all ICD models. A recent case report suggested that changes in lead parameters might be transient and may be missed. The lead may function normally as the high-voltage and pace-sense cables are covered with ETFE, which serves as the second insulating barrier. As this is a very thin layer (0.0015 inches) the reliability of this to withstand a high-energy shock is unknown. This may lead to failure of appropriate therapy for life threatening arrhythmias.

The aim of this study is to screen patients with ICD leads that potentially could have multiple different failure mechanisms, including inside-out insulation breaks, to develop a novel new algorithm and methods to detect these defects, thereby enabling physicians to prevent complications from failure of these leads.

It is hypothesized that current monitoring tools are insufficient for detecting the sometimes transient electrical failures of the Riata family of leads, and that additional device diagnostic information in combination with fluoroscopy may improve detection of electrical failures.

This will be a prospective, single-center study. Patients who consent to participate will be enrolled for up to three years.

This study offers the potential of direct benefit to the patient and indirect benefit for future users of the ICD systems. This study may identify inside-out insulation breaks and prevent impending lead failure. Additionally, analyses of the data collected as part of this study may help to develop an "electronic footprint" or pattern to remotely identify inside-out insulation breaks in all ICD leads Potential risks include exposure to radiation from a fluoroscopic exam of the lead and receiving a synchronized ICD shock.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age ≥18
* Implanted with any Medtronic Protecta® VR/DR/CRT, XT-VR/DR/CRT, Secura®, Virtuoso®, Maximo II®, Concerto® VR, Evera® or Viva® (and any future FDA-approved Medtronic ICD) device to which is attached a St. Jude Riata lead (Models 1560, 1561, 1562, 1570, 1571, 1572, 1580, 1581, 1582, 1590, 1591, 1592, 7000, 7001, 7002, 7010, 7011, 7040, 7041, 7042)
* Willing and able to sign informed consent

Exclusion Criteria:

* Age <18
* ICD that does not use a Riata lead
* Riata lead not connected to Medtronic Protecta® VR/DR/CRT, XT-VR/DR/CRT, Maximo II® Secura®, Virtuoso®, Concerto® VR, Evera® or Viva® (and any future FDA-approved Medtronic ICD) device
* Unwilling or unable to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-07; Primary Completion 2018-04 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
lead failure | 12-36 months post-enrollment
  clinical and demographic data associated with lead failure will be evaluated after 12-36 months of subject participation

CONTACTS AND LOCATIONS:
Overall Officials: Steven Zweibel, MD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

REFERENCES:
- [Background] Erkapic D, Duray GZ, Bauernfeind T, De Rosa S, Hohnloser SH. Insulation defects of thin high-voltage ICD leads: an underestimated problem? J Cardiovasc Electrophysiol. 2011 Sep;22(9):1018-22. doi: 10.1111/j.1540-8167.2011.02055.x. Epub 2011 Apr 1. PMID 21457385
- [Background] Valk S, Luijten R, Jordaens L. Insulation damage in a shock wire: an unexpected fluoroscopic image. Pacing Clin Electrophysiol. 2010 Jun 1;33(6):770-2. doi: 10.1111/j.1540-8159.2009.02664.x. Epub 2010 Jan 12. PMID 20070544